CLINICAL TRIAL: NCT01529281
Title: Exercise-induced Muscle Damage is Reduced in Resistance Trained Athletes by Branch Chain Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Northumbria_How_BCAA
Record Dates: First submitted 2012-02-02; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Exercise-induced Muscle Damage
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCAA (Experimental): Branched chain amino acid
  Interventions: Dietary Supplement: Branch Chain Amino Acid (BCAA)
- Asparmate (Placebo Comparator): Placebo control containing no protein or carbohydrate
  Interventions: Dietary Supplement: Placebo - asparmate

INTERVENTIONS:
Dietary Supplement: Branch Chain Amino Acid (BCAA) — Supplementation lasted for a total of 12 days; this was based on previous research showing a positive with BCAA supplementation on markers of muscle damage. Participants ingested 10 g, twice per day (morning and evening) of BCAA . The BCAA supplement contained a ratio of 2:1:1 (leucine, isoleucine and valine, respectively). The BCAA was in powder form where each serving was mixed with ~300 ml of water.
  Arms: BCAA
Dietary Supplement: Placebo - asparmate — Supplementation lasted for a total of 12 days. Participants ingested an equivalent looking volume to 10 g of BCAA, twice per day (morning and evening) of placebo (aspartame based artificial sweetener). The BCAA supplement contained a ratio of 2:1:1 (leucine, isoleucine and valine, respectively). The artificial sweetener was in powder form where each serving was mixed with ~300 ml of water.
  Arms: Asparmate

SUMMARY:
It is well documented that exercise-induced muscle damage (EIMD) decreases muscle function and causes severe soreness and discomfort. Branched-chain amino acid (BCAA) supplementation has been shown to increase protein synthesis and decrease muscle protein breakdown, however, the effects of BCAAs on recovery from EIMD are unknown. Thus, the aim of this study was to examine the effects of a BCAA supplement on markers of muscle damage.

ELIGIBILITY:
Inclusion Criteria:

- Resistance trained males

Exclusion Criteria:

- Muscular skeletal disorders

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary contraction | pre exercise, 24 h, 48 h, 72 h, 96 h post-exercise
  Isometric MVC of the participants' dominant knee extensors was assessed using a strain gauge. MVCs were performed for 3 s with a 60 s rest between each repetition.

SECONDARY OUTCOMES:
Limb girths | pre-exercise, 24h, 48h, 72h, 96h
  Mid-thigh and calf circumference was assessed as a measure of limb swelling using an anthropometric tape measure. Both measures were obtained with the participant in a standing position.
Vertical jump | pre-exercise, 24h, 48h, 72h, 96h
  Vertical jump (VJ) performance was assessed using the Vertec instrument. Participants performed a counter movement jump.
Creatine kinase | pre-exercise, 24h, 48h, 72h, 96h
  Plasma CK was determined from an earlobe capillary blood sample. The sample (30 microlitres) was analysed immediately using an automated, dry slide photospectrometer.
Muscle soreness | pre-exercise, 24h, 48h, 72h, 96h
  Muscle soreness - Participants were asked to perform and hold a squat (90° knee angle) whilst they rated their perceived muscle soreness on a 200 mm visual analogue scale. The scale consisted of a line from 0 mm (no pain) to 200 mm (unbearably painful).

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, PhD, Principal Investigator — Northumbria University

REFERENCES:
- [Derived] Howatson G, Hoad M, Goodall S, Tallent J, Bell PG, French DN. Exercise-induced muscle damage is reduced in resistance-trained males by branched chain amino acids: a randomized, double-blind, placebo controlled study. J Int Soc Sports Nutr. 2012 Jul 12;9:20. doi: 10.1186/1550-2783-9-20. eCollection 2012. PMID 22569039